CLINICAL TRIAL: NCT00609778
Title: A Comparison of Conventional Adult Out-of-hospital Cardiopulmonary Resuscitation Against a Concept With Mechanical Chest Compressions and Simultaneous Defibrillation
Brief Title: A Comparison of Conventional Adult Out-of-hospital Cardiopulmonary Resuscitation Against a Concept With Mechanical Chest Compressions and Simultaneous Defibrillation - LINC Study
Acronym: LINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jolife AB (Industry)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jolife 10-0
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2011-06

CONDITIONS: Cardiovascular Diseases
Keywords: CPR; Mechanical; Manual; Survival; ROSC
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1:Mechanical CPR with LUCAS (Experimental): A Mechanical device that provides chest compressions
  Interventions: Device: LUCAS
- 2 Manual CPR (Active Comparator): Manual chest compressions
  Interventions: Other: Conventional manual resuscitation method

INTERVENTIONS:
Device: LUCAS — Mechanical chest compression
  Arms: 1:Mechanical CPR with LUCAS
Other: Conventional manual resuscitation method — Manual compression
  Arms: 2 Manual CPR

SUMMARY:
The primary objective is to show superiority in survival of the modified method with the LUCAS Chest Compression System, compared to the conventional manual resuscitation method in patients suffering from out of hospital sudden cardiac arrest.

DETAILED DESCRIPTION:
Every year 300 000 to 400 000 people suffer from sudden cardiac arrest outside of the hospital in Europe. Only 5 - 7 % of these patients survive and are discharged from hospital. In spite of massive education, research and new methods the survival rate has not improved. In the latest international guidelines for CPR, published in 2005, there is a strong emphasis on chest compressions with as little interruptions as possible. Manual chest compressions during CPR result in only 20-30% of normal blood flow and are difficult to perform for a long period of time. Mechanical chest compressions with the LUCAS device have shown increased blood flow in experimental studies. Defibrillation during ongoing mechanical compressions is a new method of treatment that showed promising results in increased short time survival in out of hospital cardiac arrest in a recently completed pilot study.

The LINC trial is a prospective randomised multicenter study where LUCAS according to a concept will be used with simultaneous defibrillation compared to manual chest compressions according to 2005 guidelines for advanced CPR. The study will be conducted in first tier systems, where LUCAS always will be placed in the first arriving ambulance.

ELIGIBILITY:
Inclusion Criteria:

* Unexpected adult out-of-hospital cardiac arrest where an attempt of resuscitation is considered appropriate.

Exclusion Criteria:

* Traumatic cardiac arrest, including hanging
* Age believed to be less than 18 years (no upper limit)
* Known pregnancy
* Defibrillated before LUCAS Chest Compressions System arrives at scene
* Patients body size not fitting the LUCAS Chest Compression System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Four hour survival from successful restoration of spontaneous circulation. | Four hours survival

SECONDARY OUTCOMES:
ROSC, Arrival to the emergency room with ROSC. Survival in hospital,Survival to hospital discharge Survival 1 and 6 months ( without severe neurological impairmen (CPC 1 or 2). | Restoration of ROSC, Arrival to emergency room with ROSC, Survival to discharge from ICU, Survival to hospital discharge, Survival one and six months after SCA

CONTACTS AND LOCATIONS:
Locations (6):
- Stichting RAVU EMS, Utrecht, Netherlands
- Sweden (4):
  - Kamber, Skåne, Malmo, Skåne County
  - Gävle EMS, Gävle
  - Uppsala EMS, Uppsala
  - Västerås EMS, Västerås
- NHS, South Western Ambulance Service Trust (SWAST), Bournemouth, Poole & Dorchester, Dorset, United Kingdom

REFERENCES:
- [Derived] Rubertsson S, Lindgren E, Smekal D, Ostlund O, Silfverstolpe J, Lichtveld RA, Boomars R, Bruins W, Ahlstedt B, Skoog G, Kastberg R, Halliwell D, Box M, Herlitz J, Karlsten R. Per-Protocol and Pre-Defined population analysis of the LINC study. Resuscitation. 2015 Nov;96:92-9. doi: 10.1016/j.resuscitation.2015.07.008. Epub 2015 Aug 3. PMID 26247144
- [Derived] Rubertsson S, Lindgren E, Smekal D, Ostlund O, Silfverstolpe J, Lichtveld RA, Boomars R, Ahlstedt B, Skoog G, Kastberg R, Halliwell D, Box M, Herlitz J, Karlsten R. Mechanical chest compressions and simultaneous defibrillation vs conventional cardiopulmonary resuscitation in out-of-hospital cardiac arrest: the LINC randomized trial. JAMA. 2014 Jan 1;311(1):53-61. doi: 10.1001/jama.2013.282538. PMID 24240611
- [Derived] Rubertsson S, Silfverstolpe J, Rehn L, Nyman T, Lichtveld R, Boomars R, Bruins W, Ahlstedt B, Puggioli H, Lindgren E, Smekal D, Skoog G, Kastberg R, Lindblad A, Halliwell D, Box M, Arnwald F, Hardig BM, Chamberlain D, Herlitz J, Karlsten R. The study protocol for the LINC (LUCAS in cardiac arrest) study: a study comparing conventional adult out-of-hospital cardiopulmonary resuscitation with a concept with mechanical chest compressions and simultaneous defibrillation. Scand J Trauma Resusc Emerg Med. 2013 Jan 25;21:5. doi: 10.1186/1757-7241-21-5. PMID 23351178